CLINICAL TRIAL: NCT07184827
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of U101 Oral Capsules in the Prevention of Uncomplicated Recurrent Urinary Tract Infections (rUTIs) in Women
Brief Title: Evaluate the Efficacy and Safety of U101 Oral Capsules in the Prevention of Uncomplicated rUTIs in Women
Acronym: U101
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TCM Biotech International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TCMU101-001
Record Dates: First submitted 2025-08-05; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Urinary Tract Infections in Women
Keywords: recurrent urinary tract infections; recurrent urinary tract infections in women; rUTI; UTI; rUTIs; UTIs; pentosan polysulfate sodium; PPS; Glycosaminoglycan; Glycosaminoglycans; GAG; GAGs
MeSH Terms: conditions — Urinary Tract Infections | interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): One capsule of Placebo will be administered orally three times per day (TID) for 8 weeks followed by one capsule of placebo twice per day (BID) for 16 weeks.
  Interventions: Other: Placebo
- U101 (Experimental): One capsule (100 mg) of U101 will be administered orally three times per day (TID) for 8 weeks followed by one capsule of U101 twice per day (BID) for 16 weeks.
  Interventions: Drug: U101

INTERVENTIONS:
Drug: U101 — One capsule (100 mg) of U101 will be administered orally three times per day (TID) for 8 weeks followed by one capsule of U101 twice per day (BID) for 16 weeks.
  Other Names: pentosan polysulfate sodium (PPS)
  Arms: U101
Other: Placebo — One capsule of Placebo will be administered orally three times per day (TID) for 8 weeks followed by one capsule of placebo twice per day (BID) for 16 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug U101 works to prevent recurrent urinary tract infection (rUTI) in women (≥ 20 and < 76 years old) with a medical history. It will also investigate the safety and the impact on the Quality of Life improvement of drug U101. The main questions it aims to answer are:

* Does the drug prevent or decrease the recurrence of urinary tract infection (UTI) during the 24-week treatment?
* Will the Quality of Life be improved during the 24-week treatment?
* What medical problems do participants have when taking drug U101?

Researchers will compare drug U101 to a placebo (a look-alike substance that contains no drug) to see if drug U101 works to prevent rUTI.

Participants will:

* Orally take drug U101 or placebo every day for 24 weeks in the main study, three times per day (TID) for 8 weeks and twice per day (BID) for 16 weeks.
* Visit the site once every 4 weeks for checkups and tests during the main study.
* be asked to enroll in extensional study (the open-label extension (OLE) with drug U101 treatment or the Safety Follow-Up Visits with no investigational product treatment) for 24 weeks after they complete the 24-week main study.
* Visit the site when the suspected UTI occurred during the main study or the extension study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 3 study evaluating the efficacy and safety of U101 versus placebo in women with recurrent urinary tract infections (UTIs).

The study will be conducted primarily on an outpatient basis and consist of (1) a Screening Period, (2) a Main Study (24 weeks), and (3) an optional Open-Label Extension (OLE) program/Follow-Up Period (total 24 weeks). The study plans to enroll a total of 348 participants.

Female participants (≥ 20 and < 76 years old) who have experienced rUTIs (defined as ≥ 2 UTI events in a 6-month period or ≥ 3 UTI events in a 12-month period) but confirmed resolved infection before randomization will be the potential candidates to enroll in this study.

During the screening period, patients with a history of rUTIs who present at the study sites will be identified. The potential participants will proceed with other study-specific activities to confirm their eligibility. Once confirmed, participants will be stratified based on their menopausal status (Yes/No) and study site then randomized into the main study in a 1:1 ratio to receive U101 or matching placebo.

During the main study, one capsule (100 mg) of U101 or matching placebo will be administered orally three times per day (TID) for 8 weeks followed by one capsule of U101 or matching placebo twice per day (BID) for 16 weeks. The total study duration will be 24 weeks and participants will be required to attend site visits every 4 weeks (routine visits).

If participants develop symptoms or have a positive urinalysis result suggestive of a UTI at any time after receiving the first dose of study medication during the main study and the OLE/Follow-up period, they are instructed to contact the study staff to arrange for a special visit for examination (suspected UTI visit). If the investigator suspects a UTI recurrence and prescribes systematic antibiotics as a result, the study medication will be interrupted. After the resolution of the infection, the study medication will be reintroduced again on a TID dosing schedule.

Participants will be offered to enroll in the open-label extension (OLE) program or enter the Follow-Up Visits after they complete the 24-week main study.

The purpose of the OLE is to collect additional safety and efficacy data. Eligible participants and the investigators will decide whether the participants should receive U101 treatment (TID for 8 weeks followed by BID for 16 weeks) or enter the long-term follow-up period without any treatment. To receive U101 treatment during the OLE, participants must experience at least 1 UTI episode during the 24-week main study. The OLE will last for 24 weeks and all participants will be scheduled for two visits at Week 8 and Week 24. The OLE may be terminated contingent on the primary analysis results of the main study.

Participants who are not eligible for or who choose not to receive U101 will enter the long-term safety follow-up. This Follow-up period has the same visit schedules (at Week 8 and Week 24) as the OLE; however, no treatment will be administered.

The primary analysis will be conducted at the end of the 24-week main study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed informed consent form.
2. Non-pregnant, non-nursing females ≥ 20 and < 76 years old.
3. Having a history of ≥ 2 UTI events during the preceding 6 months or ≥ 3 UTI events during the preceding 12 months (including any UTI event that occurs on the date of ICF signing). At least one of the previous UTI events must have microbiologic evidence (e.g., per the investigator's judgment based on urine culture results).
4. The last urine culture (including those conducted for suspected UTI event or retest) before the randomization has to be negative.
5. Having a negative urinalysis result and no symptoms suggestive of a UTI on the day of randomization.

Exclusion Criteria:

1. Females who are pregnant, nursing, have a desire for pregnancy or have a positive pregnancy test at screening.
2. Women of childbearing potential who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy for the entire study period (use of spermicide is prohibited). Women of childbearing potential are defined as premenopausal females capable of becoming pregnant.
3. Serum aspartate transaminase (AST), serum alanine transaminase (ALT) and serum total bilirubin > 1.5 x upper limit of normal (ULN).
4. Serum creatinine > 1.5 x ULN.
5. Prothrombin time (PT) or INR > 1.2 x ULN.
6. Platelet counts < 100,000/μL.
7. Serum vitamin D level < 11 ng/mL.
8. HbA1c > 8.0%.
9. Positive test for hepatitis B (both HBsAg and HBeAg), hepatitis C (anti-HCV antibody) or HIV (anti-HIV antibody).
10. Symptoms suggestive of a systemic inflammatory response (fever > 38℃ or WBC count > 12,000) at the screening.
11. A major functional or anatomical abnormality of the urogenital tract (e.g., renal cell carcinoma, outlet obstruction, etc.).
12. Diagnosis of pelvic organ prolapse ≥ grade 2 (according to pelvic organ prolapse quantification POP-Q classification) without any treatment within 6 months of the screening visit.
13. Diagnosis of complicated UTIs within 6 months of the screening visit.
14. Residual urine volume > 100 mL within a month of the screening visit.
15. History of interstitial cystitis, pelvic inflammatory disease, or chronic pelvic pain syndrome.
16. Having any of the following procedures within a week of the screening: urinary catheterization (e.g., Foley catheter), ureteral stent, percutaneous nephrostomy, or cystostomy.
17. Intravesical instillation of hyaluronic acid within 6 months of the screening visit.
18. Treatment with pentosan polysulfate sodium (PPS) within 6 months of the screening visit.
19. Use of antibiotic prophylaxis for rUTI within a month of the screening visit.
20. Use of local hormone therapy (cream, gel, insert, ring, or tablets) in urogenital areas within a month of the screening.
21. Any history of thrombocytopenia, hemophilia, or bladder cancer; history of endoscopy-confirmed gastrointestinal ulcers within 3 years prior to randomization.
22. Active malignancy (under intensive cancer treatment or considered in progression) or a history of any malignancy involving the pelvic cavity within 5 years prior to randomization, with the exception of adequately treated basal cell carcinoma and cervical cancer in-situ. Subjects in stable condition will be evaluated and discussed individually with the investigator.
23. Immunocompromised or history of organ transplant.
24. History of allergies to pentosan polysulfate sodium.
25. Having planned major surgery within 24 weeks after the study.
26. Participation in any interventional clinical trial within 30 days of the screening visit.
27. Other significant medical problem(s) or intercurrent acute illness(es) that in the opinion of the Investigators, would make participation in the study unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objective.
28. Subjects who are illiterate.
29. Subjects having a family history of macular degeneration or having been diagnosed with macular degeneration (except for those with asymptomatic age-related macular degeneration) .

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects without UTI recurrence during the 24-week main study period | The primary analysis will be performed at the end of the 24-week main study
  To demonstrate the efficacy of U101 in preventing recurrent urinary tract infections (rUTIs) in women

SECONDARY OUTCOMES:
Time to the first UTI episode during the main study period | This analysis will be performed at the end of the 24-week main study
  To evaluate the specified time period of rUTI prevention after enrollment
Percentage of subjects with ≤ 1 UTI episode during the main study period | This analysis will be performed at the end of the 24-week main study
  To evaluate the percentage of rUTI ≤ 1 episode after enrollment
Average number of time-normalized UTI episodes per 4 weeks during the main study period | This analysis will be performed at the end of the 24-week main study
  To evaluate the decrease in UTI recurrence after enrollment
Quality of Life assessment: Daily Activities Interference during the main study period | This analysis will be performed at the end of the 24-week main study
  Subject self-assessment questionnaire to evaluate the degree to which daily activities are affected. Measured on a 0-4 ordinal scale, with higher scores indicating greater interference.
Quality of Life assessment: Pain Intensity during the main study period | This analysis will be performed at the end of the 24-week main study
  Evaluated using a 0-10 Numerical Rating Scale (NRS), with higher scores indicating greater pain intensity.
Quality of Life assessment: Overall Health Status during the main study period | This analysis will be performed at the end of the 24-week main study
  Evaluated using a 0-10 Numerical Rating Scale (NRS), with higher scores indicating greater pain intensity.
Quality of Life assessment: Sexual Wellbeing during the main study period(Optional) | This analysis will be performed at the end of the 24-week main study
  Evaluated on a 1-5 ordinal scale, with higher scores indicating greater willingness, symptom severity, or satisfaction. It is optional.
Quality of Life assessment: UTI questionnaires during the main study period | This analysis will be performed at the end of the 24-week main study
  Two subject self-assessment questionnaires will be used to evaluate the participants' symptom presentation during infection.
  The urinary tract infection(UTI) questionnaire is designed to evaluate the degree of symptom-related burden associated with UTI. Most items are rated on a 0-4 ordinal scale, with higher scores indicating greater symptom burden.
Treatment-emergent adverse events (TEAE), and all AE and serious adverse events (SAE) incidence rates to evaluate the safety and tolerability, during the main study period | This analysis will be performed at the end of the 24-week main study (ongoing AE/SAE will be followed up for 14 days after the subjects complete the 24-week treatment and will be included in the primary analysis)
  Adverse events will be graded according to the criteria of NCI CTCAE v5.0 and coded to the preferred term (PT) and system organ class (SOC) using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) system.
  For each treatment arm, AE incidence rates will be summarized with frequency and percentage by MedDRA SOC and preferred term. It will also be summarized by severity and relationship to the study drug.
Safety Laboratory Assessments: Hematology Abnormalities during the main study period | This analysis will be performed at the end of the 24-week main study
  Number of participants with abnormal hematology results (e.g., complete blood count parameters such as hemoglobin, white blood cells, platelets) as assessed using standard laboratory methods. Abnormalities will be graded according to NCI CTCAE v5.0.
Safety Laboratory Assessments: Serum Chemistry Abnormalities during the main study period | This analysis will be performed at the end of the 24-week main study
  Number of participants with abnormal serum chemistry results (e.g., liver function tests, kidney function tests, electrolytes) assessed using standard laboratory methods. Graded according to NCI CTCAE v5.0.
Safety Laboratory Assessments: Coagulation Abnormalities during the main study period | This analysis will be performed at the end of the 24-week main study
  Number of participants with abnormal coagulation parameters (e.g., PT, aPTT, INR) assessed using standard laboratory methods. Graded according to NCI CTCAE v5.0.
Safety Laboratory Assessments: Urinalysis Abnormalities during the main study period | This analysis will be performed at the end of the 24-week main study
  Number of participants with abnormal urinalysis results (e.g., protein, glucose, blood) assessed using standard laboratory methods. Graded according to NCI CTCAE v5.0.
Vital signs (Blood pressure) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the systolic and diastolic blood pressure.
Vital signs (Pulse rate) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the pulse rate.
Vital signs (Respiratory rate) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the respiratory rate.
Vital signs (Body temperature) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the body temperature.
Vital signs (Weight) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the weight.
Physical examination (Height) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the height.
Physical examination (Skin) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the skin.
Physical examination (Neck) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the neck.
Physical examination (Eyes) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the eyes.
Physical examination (Ears) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the ears.
Physical examination (Nose) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the nose.
Physical examination (Throat) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the throat.
Physical examination (Breast) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the breast.
Physical examination (Lungs) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the lungs.
Physical examination (Heart) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the heart.
Physical examination (Abdomen) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the abdomen.
Physical examination (Back) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the back.
Physical examination (Lymph Nodes) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the lymph nodes.
Physical examination (Extremities) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the extremities.
Physical examination (Nervous System) during the main study period | This analysis will be performed at the end of the 24-week main study
  Clinically significant changes in the nervous system.

CONTACTS AND LOCATIONS:
Overall Officials: En Meng, MD, Principal Investigator — Tri-Service General Hospital
Locations (13):
- Taiwan (13):
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital, Taipei Branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital (TSGH), Taipei
  - Chang Gung Memorial Hospital, Linkuo Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No